CLINICAL TRIAL: NCT04144751
Title: Blood Collection Sub-Study of Exact Sciences Protocol 2019-01: "Clinical Validation of an Optimized Multi-Target Stool DNA (Mt-sDNA 2.0) Test, For Colorectal Cancer Screening BLUE-C"
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-01B
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: Blood Draw
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples may be used for evaluating performance of biomarkers for feasibility and assay development. Sample may be stored for up to 20 years. These blood samples will be de-identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects Enrolled in 2019-01 BLUE-C: Subjects will be men and women, 40 years of age or older, who enroll in Exact Sciences Protocol 2019-01 BLUE-C. Subjects will provide a blood sample at time of enrollment.
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Subjects participating in the study will have blood drawn at enrollment.

SUMMARY:
The primary objective of this sub-study, 2019-01B, is to collect blood specimens for research use in the development and validation of a blood-based test for colorectal cancer (CRC).

DETAILED DESCRIPTION:
Subjects who consent to enroll in Exact Sciences Protocol 2019-01 BLUE-C, will be invited to participate in this sub-study. Subjects enrolled in the Exact Sciences Protocol 2019-01 BLUE-C, who provide written informed consent to participate in this sub-study, will have a blood sample collected at enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is currently enrolled in Exact Sciences Protocol 2019-01 BLUE-C.
2. Subject is willing and able to provide a blood sample.
3. Subject is willing and able to sign informed consent.

Exclusion Criteria:

1. Subject has any condition that in the opinion of the Investigator should preclude participation in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be men and women, 40 years of age or older, who enroll in Exact Sciences Protocol 2019-01 BLUE-C. Up to 24,000 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 23494 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Blood-based biomarkers associated with genetic and epigenetic alterations. | Point in time blood collection (1 day) at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Imperiale, MD, Principal Investigator — Indiana University
Locations (193):
- United States (193):
  - Parkway Medical Center, Birmingham, Alabama
  - Summit Internal Medicine, PC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - G & L Research, Foley, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - East View Medical Research, LLC, Mobile, Alabama
  - GI Associates of West Alabama, P.C, Tuscaloosa, Alabama
  - Mayo Clinic - AZ, Phoenix, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Southern Arizona VA Health Care System (SAVAHCS), Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Arkansas Gastroenterology, P.A., North Little Rock, Arkansas
  - Fomat Medical Research, Camarillo, California
  - Alliance Research Institute, Canoga Park, California
  - GW Research Inc, Chula Vista, California
  - Paragon Rx Clinical, Inc., Garden Grove, California
  - United Medical Doctors, Irvine, California
  - Prime Care Clinical Research Center, Laguna Hills, California
  - Gastro Care Institute, Lancaster, California
  - Facey Medical Foundation, Mission Hills, California
  - Knowledge Research Center, Orange, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Palo Alto Veterans Institute for Research, Palo Alto, California
  - SDG Clinical Research, San Diego, California
  - San Jose Gastroenterology, San Jose, California
  - Paragon Rx Clinical, Inc. - Santa Ana, Santa Ana, California
  - Sansum Clinic, Santa Barbara, California
  - Unison Clinical Trials, Sherman Oaks, California
  - Millennium Clinical Trials, Thousand Oaks, California
  - Dream Team Clinical Research, Upland, California
  - New West Physicians, Golden, Colorado
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Yale University, New Haven, Connecticut
  - Cornerstone Research Institute, Altamonte Springs, Florida
  - Vanguard Clinical Research, Fort Myers, Florida
  - SIMED Health Research, Gainesville, Florida
  - Westside Center of Clinical Research, Jacksonville, Florida
  - Shands Jacksonville Medical Center, Inc - University of Florida Health, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Wr-Msra, Llc, Lake City, Florida
  - Alliance Medical Research, Lighthouse PT, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Next Phase Research Alliance, Miami, Florida
  - Research Associates of South Florida, LLC, Miami, Florida
  - Gastro Health Research, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Sarkis Clinical Trials, Ocala, Florida
  - Imic, Inc., Palmetto Bay, Florida
  - Family Medical Specialists of Florida, PLC, Plant City, Florida
  - Alternative Solutions, LLC, St. Petersburg, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Clinical Trials of Tampa, Tampa, Florida
  - Summit Clinical Research, LLC, Athens, Georgia
  - Augusta University, Augusta, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Infinite Clinical Trials, Morrow, Georgia
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Christie Clinic, Champaign, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - GI Partners of IL / Avicenna, Downers Grove, Illinois
  - Edward Hines Jr. VA Hospital, Hines, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Deaconess Clinic, Inc., Newburgh, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - PMG Research, Ames, Iowa
  - University of Iowa, Iowa City, Iowa
  - The Iowa Clinic, P.C., West Des Moines, Iowa
  - Digestive Health Center of the Four States, LLC, Galena, Kansas
  - Hutchinson Clinic, Hutchinson, Kansas
  - Ascension Via Christi Hospitals Wichita, Inc, Wichita, Kansas
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Horizon Research Group of Opelousas, LLC, Eunice, Louisiana
  - Houma Digestive Health Specialists-CroNOLA, Houma, Louisiana
  - Combined Gastro Research. LLC, Lafayette, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - New Orleans Research Institute, Metairie, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Louisiana Research Center; Gastrointestinal Associates, Shreveport, Louisiana
  - Clinical Trials of America, LLC, West Monroe, Louisiana
  - Gastro Health Research, Annapolis, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - Harvard, Boston, Massachusetts
  - IQVIA RDS, Inc., Cambridge, Massachusetts
  - Digestive Health Specialists, PC, Chelmsford, Massachusetts
  - NECCR PrimaCare Research, LLC, Fall River, Massachusetts
  - University of Massachusetts - Worcester, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Oakland Medical Research, Troy, Michigan
  - Center for Digestive Health Research, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research LLC (STAR), Jackson, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Methodist Physicians Clinic / CCT Research, Fremont, Nebraska
  - CHI Nebraska, Omaha, Nebraska
  - University of Nevada, Las Vegas, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Digestive Health Associates, Reno, Nevada
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Allied Health Clinical Research Organization, LLC, West Long Branch, New Jersey
  - United Health Services Hospitals, Inc., Binghamton, New York
  - VA NY Harbor HCS- Brooklyn Campus, Brooklyn, New York
  - Sing Chan, MD, Flushing, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - DiGiovanna Institute for Medical Education & Research, North Massapequa, New York
  - Digestive Health Partners, PA, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Department of Family Medicine Research, Charlotte, North Carolina
  - Javara, Charlotte, North Carolina
  - Coastal Research Institute, LLC, Fayetteville, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Clinical Trials of America, LLC, Mount Airy, North Carolina
  - Coastal Carolina Health Care, P.A, New Bern, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Great Lakes Medical Research LLC, Beachwood, Ohio
  - Gastro Health Research, Cincinnati, Ohio
  - Hightop Medical Research Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - META Medical Research Institute, LLC, Dayton, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Paramount Medical Research and Consulting, LLC, Middleburg Heights, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Comprehensive Internal Medicine, Inc, Wooster, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - SSM Health Medical Group/Hightower Clinical, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Great Lakes Medical Research, LLC, Harrisburg, Pennsylvania
  - Richard M. Kastelic, M.D., and Associates, P.C., Johnstown, Pennsylvania
  - Regional GI, Lancaster, Pennsylvania
  - Thomas Jefferson University Philadelphia, Philadelphia, Pennsylvania
  - Care Access Research, Pottsville, Pottsville, Pennsylvania
  - Ralph H. Johnson VAMC, Charleston, South Carolina
  - Pharmacorp Clinical Trials, Inc., Charleston, South Carolina
  - Invocare Medical Research & Healthcare Center, West Columbia, South Carolina
  - Rapid City Medical Center, LLP, Rapid City, South Dakota
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Clinical Research Solutions, LLC - TN, Jackson, Tennessee
  - Tri-Cities Gastroenterology, Kingsport, Tennessee
  - Great Lakes Medical Research, LLC, Union City, Tennessee
  - ARC Clinical Research at Four Points, Austin, Texas
  - Elligo Health Research Inc, Austin, Texas
  - ARC Clinical Research at William Cannon, Austin, Texas
  - Avant Research Associates, Austin, Texas
  - Mercy Family Clinic, Dallas, Texas
  - Dharma PA D/B/A Southwest Family Medicine Associates, Dallas, Texas
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
  - Houston Digestive Disease, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Fairway Medical Clinic, Houston, Texas
  - Digestive System Healthcare, Houston, Texas
  - FMC Science, LLC, Lampasas, Texas
  - Rio Grande Gastroenterology, McAllen, Texas
  - Wellness Clinical Research, McKinney, Texas
  - ARC Clinical Research at Kelly Lane, Pflugerville, Texas
  - Epic Medical Research LLC, Red Oak, Texas
  - Clinical Associates in Research Therapeutics of America, San Antonio, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - A & U Family Medicine, Sugar Land, Texas
  - Texas Gastro Consultants, Tomball, Texas
  - Progressive Clinical Research, LLC, Bountiful, Utah
  - Tanner Clinic, Layton, Utah
  - Advanced Research Institute, Ogden, Utah
  - Advanced Clinical Research, Riverton, Utah
  - Granger Medical Clinic, Riverton, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Summit Clinical Research, Petersburg, Virginia
  - Central Virginia VA Healthcare System, Richmond, Virginia
  - Virginia Gastroenterology Institute, Suffolk, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Spokane Gastroenterology, Spokane, Washington
  - Wentachee Valley Hospital, Wenatchee, Washington
  - University Physicians and Surgeons, Inc.(Marshall Health), Huntington, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study may be shared after de-identification. This may include text, tables, figures, and appendices. The study protocol and informed consent form may also be shared. Data may be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Supporting Information: Study Protocol, ICF
Time Frame: Data may be available from 2 years and ending 4 years after publication.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research.